CLINICAL TRIAL: NCT00097461
Title: Revising Employee Benefits for the Sake of Health
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 050008; 05-CC-0008
Record Dates: First submitted 2004-11-23; First posted 2004-11-24 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-04-18

CONDITIONS: Healthy
Keywords: Employee Health; Insurance Benefit; Fringe Benefit; Health Status; Socioeconomic Factors

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will explore ways in which employee benefits may be designed to improve people's health, through examining the viewpoints and preferences of low-income people. A person's health is affected not only by being able to receive health care but also by several factors such as income and education. People with lower incomes have been found to be not as healthy as those with higher incomes. While the governments of many countries in the Organization for Economic Cooperation and Development are currently working on public policy to address this topic, the likelihood is small that the United States, given its market-based economy, will do the same. However, owing to the heavy reliance in the United States on employer-sponsored health insurance, it would be useful to explore the possibility of insuring some of the measures that people can take to improve their health, and to do that through employee benefit packages. Solutions might include extended unemployment insurance, more education, job training, exercise programs, help for housing, disability insurance, and extra retirement benefits.

Adults who have a minimum of a sixth-grade reading level, have low incomes, are English speaking may be eligible for this study. For recruitment, 400 people who live and work in the Washington, D.C, area will be invited to participate, and about12 people will take part in each session. Unless people in the study participate during working hours, they will each be paid $75 at the conclusion of the session.

The study consists of one phase, in which participants will engage in a group exercise that lasts for approximately 2-1/2 hours. During that time, participants will have the chance to say what employee benefits they would choose, if the opportunity arose, to improve their health. They will first make those choices by themselves and then make choices along with other people in the group. While group members talk, the discussion will be recorded on a tape recorder. Participants will be asked to give information about themselves and their opinions but will not be asked for any information that identifies them personally, except for data needed to pay participants with a paycheck. They will also get to use a computer and will be shown how to use it, if necessary. If videotaping or photographs are done during the exercise, the investigators of the study will ask for separate signed permission to do so. Participants will be asked to respect the privacy of others in the group and to not discuss the opinions of others after leaving the session.

DETAILED DESCRIPTION:
An individual's health is affected not only by access to health care but also by a number of determinants such as income and education. Individuals with low incomes are not as healthy as those with higher incomes. Thus it seems important to explore possible avenues for improving the health of low income individuals with an eye toward ameliorating the complicated determinants of health status, aside from health insurance. Many countries in the Organization for Economic Cooperation and Development (OECD) are currently developing public policy to address this issue. In the U.S., however with its market based economy, the likelihood of adopting this public policy approach is small. Given that reality, is it possible to explore other avenues such as designing employee benefit packages with the aim of ameliorating the socio-economic determinants of health?

Objective: The goal of this project is to explore the feasibility of designing employee benefits in a manner that may improve their health, by ascertaining the perspectives and preferences of low income employees regarding employee benefits designed to ameliorate the social determinants of health. Four hundred male and female low-income individuals recruited from clinical, community, and employment settings will participate in small group exercises in which a facilitated discussion will take place using a previously tested group decision tool (CHAT: Choosing Health plans All Together) that has been modified for this project. Data will be anonymously collected regarding socio-demographic characteristics, attitudes toward health, preferences for possible employee benefits and assessment of the exercise. Group discussions will be audio-taped. Data will be analyzed quantitatively to determine preferences of employee benefits and socio-demographic factors associated with these preferences. Discussions will undergo qualitative analysis go explore the underlying reasons for participant preferences. Participants will receive $75 dollars as compensation for their participation unless they participate during working hours.

Risks and Benefits: Given the anonymous nature of the data collection we anticipate no risks other than those entailed in discussion of poor health outcomes associated with lack of insurance and low income. Participants may benefit from learning about factors that improves health status.

Outcome and Meaning to the Field: Study results will yield information about what employee benefits would be of utmost priority to low income employees. This is unique information that may contribute to efforts to find affordable strategies for ameliorating the socio-economic determinants of health for the low-income working population in the US.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Men and women who are between the ages of 18-65, and are employed with an income of up to three times the federal poverty level will be included in this study so that information can be learned about the employee benefit preferences of low-income employees.
* Minority individuals, particularly African Americans and English speaking Hispanics will be included, and will be recruited to represent one third of the study sample because of the high prevalence of minorities among the low-income population in the US.

EXCLUSION CRITERIA:

* Non-English speakers will be excluded because they will be unable to participate in the discussion that participants engage in about the reasons for their benefit choices.
* Individuals who cannot read at a 6th grade level, will be excluded because they will have difficulty reading information provided on the computer screen during the exercise.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2004-09-28; Study Completion 2017-04-18

CONTACTS AND LOCATIONS:
Overall Officials: Marion Danis, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Danis M, Biddle AK, Dorr Goold S. Insurance benefit preferences of the low-income uninsured. J Gen Intern Med. 2002 Feb;17(2):125-33. doi: 10.1046/j.1525-1497.2002.10609.x. PMID 11841528
- [Background] Danis M, Biddle AK, Goold SD. Enrollees choose priorities for Medicare. Gerontologist. 2004 Feb;44(1):58-67. doi: 10.1093/geront/44.1.58. PMID 14978321